CLINICAL TRIAL: NCT00002730
Title: PILOT STUDY OF BUTHIONINE SULFOXIMINE (BSO) IN COMBINATION WITH MELPHALAN FOR HIGH RISK NEUROBLASTOMA PATIENTS
Brief Title: Chemotherapy in Treating Children With Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CHLA-95-083; CDR0000064620 (Registry Identifier: PDQ (Physician Data Query)); NCI-T95-00920
Record Dates: First submitted 1999-11-01; First posted 2004-09-01 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Buthionine Sulfoximine; Melphalan

INTERVENTIONS:
Drug: buthionine sulfoximine
Drug: melphalan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Some tumors become resistant to chemotherapy drugs. Combining buthionine sulfoximine with chemotherapy may reduce resistance to the drug and allow more tumor cells to be killed.

PURPOSE: Phase I trial to study the effectiveness of melphalan, buthionine sulfoximine, and G-CSF in treating children with progressive neuroblastoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Describe the toxic effects of combined chemotherapy with buthionine sulfoximine (BSO) and melphalan (L-PAM) in pediatric patients with progressive neuroblastoma. II. Determine the pharmacokinetics of BSO/L-PAM in pediatric patients. III. Assess the ability of BSO to deplete glutathione by at least 90% in tumor metastatic to bone marrow, in normal marrow, and in peripheral blood lymphocytes. IV. Estimate the response rate in these patients treated with BSO/L-PAM within the confines of a pilot study.

OUTLINE: The following acronyms are used: BSO Buthionine sulfoximine, NSC-326231 L-PAM Melphalan, NSC-8806 G-CSF Granulocyte Colony-Stimulating Factor, NSC-614629 Single-Agent Chemotherapy with Drug Resistance Inhibition. L-PAM/BSO.

PROJECTED ACCRUAL: At least 18 patients will be entered to provide an adequate number of patients with marrow involvement; if the BSO dose is increased to achieve adequate GSH depletion in the marrow, an additional 12 patients will be entered. If less than 50% of patients have tumor metastatic to marrow at entry, there will be a proportional increase in the total number of patients required.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Neuroblastoma histologically confirmed at initial diagnosis or demonstration of malignant, small, round cell tumor with elevated catecholamine metabolites Refractory to conventional therapy and other higher priority therapy

PATIENT CHARACTERISTICS: Age: No greater than 21 at diagnosis Performance status: 0-2 Life expectancy: At least 2 months Hematopoietic: Cytopenias from marrow involvement eligible with study chairman approval ANC at least 1,000 Platelets at least 100,000 (transfusion independent) Counts between 70,000-100,000 allowed provided: Autologous bone marrow or peripheral stem cells available for rescue Study chairman approves entry Hemoglobin at least 8 g/dL (may transfuse) Hepatic: Bilirubin no greater than 1.5 times normal AST/ALT less than 2.5 times normal Renal: Creatinine no greater than 1.5 times normal OR Creatinine clearance or radioisotope GFR at least 70 mL/min per 1.73 square meters Pulmonary: No history of dyspnea at rest No exercise intolerance Other: No active infection requiring hospitalization No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile patients during and for 2 months after study Patients unable to receive blood products due to religious reasons may receive buthionine sulfoximine alone

PRIOR CONCURRENT THERAPY: At least 6 months since myeloablative therapy with bone marrow transplantation Recovered from toxic effects of prior therapy Biologic therapy: Not specified Chemotherapy: At least 3 weeks since chemotherapy (6 weeks since mitomycin or nitrosourea) Endocrine therapy: Not specified Radiotherapy: At least 6 weeks since radiotherapy to any extremity site or significant marrow-containing compartment At least 6 months since the following: More than 24 Gy craniospinal irradiation Total abdominopelvic plus lung irradiation Mantle plus Y-port irradiation Total-body irradiation No palliative radiotherapy to bony lesions within 1 month after entry Surgery: Not specified

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1996-06

CONTACTS AND LOCATIONS:
Overall Officials: C. Patrick Reynolds, MD, PhD, Study Chair — Children's Hospital Los Angeles
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania